CLINICAL TRIAL: NCT00211198
Title: Open Label Study of ONTAK® (Denileukin Diftitox, DAB389IL-2) to Estimate Response in Cutaneous T-Cell Lymphoma (CTCL) According to CD25 Status
Brief Title: Study of ONTAK® to Treat Cutaneous T-Cell Lymphoma (CTCL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Tufts Medical Center (Other); National Cancer Institute (NCI) (NIH); Ligand Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #33; NCT00279396 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2008-02

CONDITIONS: Lymphoma, T-Cell, Cutaneous
Keywords: Cutaneous; T-cell lymphoma; ONTAK; CD25
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell | interventions — denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ONTAK (denileukin difitox, DAB389IL-2)

SUMMARY:
The purpose of this research study is to evaluate how effective ONTAK is in the treatment of cutaneous T-cell Lymphoma (CTCL) and determine whether the presence of a type of protein called CD25 on the cancer cells makes a difference in how the body responds to the treatment.

The hypothesis is that there is no difference in response rate for patients whose tumor cells are CD25 positive or negative.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or recurrent cutaneous T-cell lymphoma (CTCL) Stage IB-IVA as defined by TNM staging.
* Pathologic proven diagnosis (cytologically confirmed) of CTCL documented in patient history.
* Preserved organ function: Creatinine and/or Liver Function levels <1.5 times institutional upper limits of normal (ULN).
* Adequate liver function as indicated by bilirubin < or equal to 1.5 times ULN, ALT < or equal to 2 times ULN, AST < or equal to 2 times ULN.
* Albumin >3.0 g/dL
* Adequate renal function as indicated by SCr < or equal to 2.5 mg/dl.
* ECOG performance status between 0-2.
* Women of childbearing potential should be screened for pregnancy prior to treatment and utilize effective contraceptive methods (e.g. barrier) during treatment period.
* Patients over the age of 18 who are willing and able to provide Informed Consent.

Exclusion Criteria:

* Pathology consistent with peripheral T-cell lymphoma.
* Stage IVB (visceral involvement with CTCL, other than lymph node involvement).
* History of Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C infection.
* Patients who are pregnant or breast feeding.
* Allergy to or have history of allergy to diphtheria toxin or IL-2.
* Previous ONTAK® usage.
* Unstable cardiovascular disease.
* Patients who have received systemic or topical antineoplastic therapy or investigational medications within past 14 days. Exception: Clear evidence of disease progression requiring immediate intervention and in the absence of ongoing toxicity from prior therapy.
* Ongoing deep vein thrombosis or a diagnosis of deep vein thrombosis less than 3 months prior to protocol enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2001-05; Primary Completion 2005-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To estimate response rates (CR + CCR + PR) according to CD25 status (CD25 positive and negative) after 4 cycles of ONTAK.

SECONDARY OUTCOMES:
Physician's Global Assessment (PGA)
Time to Event Variables - Time to response, remission, treatment failure
Response based on the CD25 status
Response based on patient demographics: stage of disease, age, sex, performance status, total dose
Number of cycles completed
6. Assess safety and tolerability of ONTAK

CONTACTS AND LOCATIONS:
Overall Officials: Francine Foss, M.D., Study Chair — Yale University
Locations (9):
- United States (9):
  - City of Hope National Medical Center, Duarte, California
  - Yale University School of Medicine, New Haven, Connecticut
  - The University of Iowa, Iowa City, Iowa
  - New England Medical Center, Boston, Massachusetts
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Francine Foss, Madeleine Duvic, Larisa Geskin, Joseph Anderson, Pierluigi Porcu, Raymond J. Hohl, Maureen Cooper, Jasmine M. Zain, John Zic, Patrica Hibberd, and Mark Acosta Efficacy and Safety of Denileukin Diftitox (Ontak®) in the Treatment of Cutaneous T-Cell Lymphoma (CTCL) According to CD25 Status. Blood (ASH Annual Meeting Abstracts), Nov 2006; 108: 2712.